CLINICAL TRIAL: NCT03183180
Title: Prevalence of Secondary Cardiac Damage in Rheumatic Fever Patients and Adherence to Penicillin Secondary Prophylaxis
Brief Title: Prevalence of Secondary Cardiac Damage in Rheumatic Fever Patients and Penicillin Secondary Prophylaxis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assuta Hospital Systems (Other)
Responsible Party: Principal Investigator, Dr. Amir Ben-Tov, Medical Director online centers, Assuta Hospital Systems
Other Study IDs: 0137-16-ASMC
Record Dates: First submitted 2017-06-07; First posted 2017-06-09 (Actual); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: Secondary Cardiac Damage in Rheumatic Fever
MeSH Terms: interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Echocardiogram — Current cardiac state will be assessed by an experienced cardiologist, including a full new Echocardiogram examination

SUMMARY:
According to American Heart Association criteria, patients who have had Rheumatic Fever (RF) should be treated with antibiotic prophylaxis. Continuous prophylaxis is recommended in patients with well-documented histories of RF and in those with evidence of rheumatic heart disease.

There is a limited data regarding adherence of patients to treatment and efficacy of treatment.

In this study, patients with RF who are older than 21 years will be collected from a computerized database of 'Maccabi Healthcare Services', one of the biggest Israeli Health Funds. Patients will be assigned to the study after obtaining informed consent.

Previous adherence to antibiotic prophylaxis will be examined according to computerized database of drugs which were issued to the patient since RF diagnosis.

Past history of cardiac involvement, including past Echocardiograms, will be collected from computerized database. In addition, the current cardiac state will be assessed by an experienced cardiologist, including a full new Echocardiogram examination.

ELIGIBILITY:
Inclusion Criteria:

- Patients older than 21 years who were diagnosed with RF (before age 18 years) according to the computerized database.

Exclusion Criteria:

* patients with other rheumatic disease diagnosed before RF diagnosis
* patients with other cardiac disease diagnosed before RF diagnosis
* patients with neoplastic disease diagnosed before RF diagnosis

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients older than 21 years who were diagnosed with RF (before age 18 years) acoording to the computerized database.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-06 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Cardiac function including vulvar involvement | 60 days
  Cardiac morphology and function measured by echocardiography

IPD SHARING:
Plan to Share IPD: Undecided